CLINICAL TRIAL: NCT04119336
Title: A Phase II Study of Nivolumab in Combination With Ixazomib, Cyclophosphamide, and Dexamethasone in Relapsed and Refractory Multiple Myeloma
Brief Title: Nivolumab, Ixazomib, Cyclophosphamide, and Dexamethasone in Relapsed/Refractory Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closure initiated by industry funding sponsor for commercial reasons.
Sponsor: Andrew Yee, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Andrew Yee, MD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-283
Record Dates: First submitted 2019-10-05; First posted 2019-10-08 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
Keywords: Refractory Multiple Myeloma; Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Nivolumab; ixazomib; Dexamethasone; Calcium Dobesilate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and Ixazomib (Experimental): - Participants will receive Nivolumab, Ixazomib, Cyclophosphamide, and Dexamethasone on a 28-day cycle.
  * Oral:
    * Ixazomib given weekly on days 1, 8, 15
    * Dexamethasone given weekly during cycle
  * Infused:
    * Nivolumab given once per cycle
    * Cyclophosphamide given on days 1, 8, 15 during cycle
  Interventions: Drug: Nivolumab; Drug: Ixazomib; Drug: Dexamethasone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Nivolumab — Given intravenously once per cycle
  Other Names: Opdivo
Drug: Ixazomib — Given orally on days 1, 8, 15.
  Other Names: Ninlaro
Drug: Dexamethasone — Given orally on days 1, 8, 15, 22
  Other Names: Decadron
Drug: Cyclophosphamide — Given intravenously on days 1, 8, 15.
  Other Names: Cytoxan

SUMMARY:
This research is being done to assess the effectiveness and safety of the combination of nivolumab with ixazomib, cyclophosphamide, and dexamethasone in relapsed and refractory multiple myeloma.

DETAILED DESCRIPTION:
This research study is a phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

* The U.S. Food and Drug Administration (FDA) has not approved nivolumab for relapsed and refractory Multiple Myeloma but it has been approved for other uses.
* The FDA has approved ixazomib and cyclophosphamide as treatment options for your disease.
* Nivolumab is a type of antibody (a protein that attaches to other cells to fight off infection and disease) that attaches to and inhibits a protein called PD-1.

  -- PD-1 is a checkpoint protein on immune cells called T cells. It normally acts as a type of "off switch" that helps keep the T cells from attacking other cells in the body. Some cancer cells have large amounts of PD-L1 which binds to PD-1 and turns off the immune system. Nivolumab inhibits PD-1 and helps take the "brake" off the immune system. The investigators' hope that nivolumab will inhibit the PD-1 protein, thus allowing your immune cells to recognize and destroy cancer cells.
* Ixazomib is a type of inhibitor that blocks a protein in your cells called a proteasome. This protein is responsible for breaking down other proteins in your cells when they need to be disposed of. By blocking the proteasome from working, a buildup of proteins will be created in the cancer cells, which may lead to cell death.
* The investigators hope that the combination of ixazomib and nivolumab with standard of care chemotherapy cyclophosphamide and dexamethasone will work together with ixazomib and nivolumab to treat multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated relapsed and refractory multiple myeloma per International Myeloma Working Group consensus criteria (Rajkumar et al., 2011).
* Patients must have received at least three prior lines of therapy, including an immunomodulatory drug (e.g. lenalidomide, pomalidomide), a proteasome inhibitor (e.g. bortezomib, carfilzomib), and anti-CD38 monoclonal antibody (e.g. daratumumab)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (see Appendix A).
* Age ≥ 18 years
* All laboratory assessments for eligibility should be performed within 21 days of initiation of protocol therapy unless otherwise specified.
* Measurable disease of multiple myeloma as defined by at least one of the following (IgD and IgA with monoclonal protein < 0.5 g/dL may be permitted after discussion with PI):

  * Serum monoclonal protein ≥ 0.5 g/dL (or quantitative IgA ≥ 1000 mg/dL), or
  * ≥ 200 mg of monoclonal protein in the urine on 24-hour urine protein electrophoresis, and/or
  * Serum free light chain ≥ 100 mg/L (10 mg/dL) and abnormal serum free kappa to serum free kappa light chain ratio
* ANC ≥ 1000/μL. G-CSF is not permitted within 14 days of screening.
* Platelet count ≥ 75,000/µL. Platelet transfusions are not permitted within 7 days of screening.
* Hemoglobin ≥ 8 g/dL. Red blood cell transfusions are permitted to meet eligibility criteria.
* Calculated creatinine clearance of ≥ 30 mL/min according to Cockroft-Gault equation.
* Adequate hepatic function, as evidenced by each of the following:

  * Serum aspartate transaminase (ALT) and/or aspartate transaminase (AST) values < 3 × the institutional upper limit of normal (ULN).
  * Serum bilirubin values < 1.5 mg/dL. Patients with elevated bilirubin due to Gilbert's syndrome may be permitted with PI approval.
* Able to swallow capsules whole (ixazomib capsules should not be crushed, dissolved or broken).
* Women of childbearing potential (WOCBP)* must agree to follow instructions for methods of contraception for the duration of study treatment with nivolumab and for five months after the last dose of study treatment. If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through five months after the last dose of study drug OR agree to practice true abstinence when it in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

  -- Women of child bearing potential are women who are not postmenopausal for at least one year and who are not surgically sterile.
* Males who are sexually active (even if surgically sterilized, i.e. vasectomy) with WOBCP must agree to follow instructions for methods of contraception for the duration of study treatment with nivolumab and 7 months after the last dose of study treatment. Agree to practice effective barrier contraception during the entire study treatment period and through 7 months after the last dose of study drug, or agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Patient has given voluntary, signed written informed consent before performance of any study-related procedure that is not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care

Exclusion Criteria:

* Prior therapy with ixazomib
* Prior therapy with any anti-PD1 antibody (e.g. nivolumab, pembrolizumab) or anti-PDL1 antibody (e.g. atezolizumab, avelumab, durvalumab)
* Participants who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) or with monoclonal antibodies 3 weeks of C1D1 or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier. Patients may have received dexamethasone within 2 weeks prior to C1D1.
* Participation in other clinical trials, including those with other investigational agents, within five half-lives prior to C1D1and throughout the duration of this trial. Prior treatment with an investigational agent within five half lives prior to C1D1 may be permitted after discussion with the PI.
* Concomitant high-dose corticosteroid use except chronic steroids (maximum dose 10 mg/day prednisone equivalent) if they are being given for disorders other than myeloma, e.g. adrenal insufficiency, rheumatoid arthritis, etc.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period (within 21 days of C1D1).
* Prior history of malignancies, other than MM, unless the patient has been free of the disease for ≥ 3 years. Exceptions include the following if the patient has undergone complete resection:

  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Ductal carcinoma in situ of the breast
  * Incidental histologic finding of prostate cancer (T1a or T1b)
* Patients with another malignancy undergoing active treatment with the exception of non-melanoma skin cancer or in situ cervical cancer.
* Patients with plasma cell leukemia, POEMS syndrome, or amyloidosis are excluded from this trial.
* HIV infection.
* Active hepatitis B infection or active hepatitis C infection. Participants who have prior hepatitis C infection and who have received an antiviral treatment and show no detectable viral RNA for 6 months prior to screening are eligible.
* Peripheral neuropathy ≥ grade 2 despite supportive therapy.
* Prior allogeneic stem cell transplant within five years prior to study registration. Patients who have had an allogeneic stem cell transplant within five years prior to study registration may participate as long as there are no symptoms of graft versus host disease.
* Patient has a history of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory, or inflammatory illness that could preclude study participation, pose an undue medical hazard, or interfere with the interpretation of the study results, including, but not limited to, patients with congestive heart failure (New York Heart Association [NYHA] Class 3 or 4); unstable angina; cardiac arrhythmia; recent (within the preceding 6 months) myocardial infarction or stroke; hypertension requiring > 2 medications for adequate control; diabetes mellitus with > 2 episodes of ketoacidosis in the preceding 12 months; or chronic obstructive pulmonary disease (COPD) requiring > 2 hospitalizations in the preceding 12 months.

3.2.15 Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune pneumonitis, autoimmune vasculitis (e.g., Wegener's granulomatosis) and motor neuropathy considered of autoimmune origin (e.g. Guillain-Barré syndrome and myasthenia gravis). Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

* Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
* Major surgery within 14 days prior to study registration.
* Central nervous system involvement.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days prior to study registration
* Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort within 14 days prior to C1D1.
* Receipt of a live or attenuated vaccine within 30 days of C1D1.
* Any serious medical of psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any study medications, their analogs, or excipients in the various formulations of any agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Yee, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation
URL: http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab and Ixazomib: - Participants will receive Nivolumab, Ixazomib, Cyclophosphamide, and Dexamethasone on a 28-day cycle.
  * Oral:
    * Ixazomib given weekly on days 1, 8, 15
    * Dexamethasone given weekly during cycle
  * Infused:
    * Nivolumab given once per cycle
    * Cyclophosphamide given on days 1, 8, 15 during cycle
  Nivolumab: Given intravenously once per cycle
  Ixazomib: Given orally on days 1, 8, 15.
  Dexamethasone: Given orally on days 1, 8, 15, 22
  Cyclophosphamide: Given intravenously on days 1, 8, 15.
Period: Overall Study
Arm/Group | Nivolumab and Ixazomib
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab and Ixazomib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as percentage of participants with complete response (CR) and partial response (PR) per International Myeloma Working Group (IMWG) criteria below.
  * CR = Negative immunofixation on serum and urine; disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow
  * Stringent CR = Above definition plus normal FLC ration and absence of clonal cells in bone marrow by IHC or 2-4 color flow cytometry
  * PR = At least 50% reduction of serum M-protein and reduction in 24 urinary M-protein by at least 90% or to <200 mg/24 h. If serum and urine M-protein unmeasurable, require at least 50% decrease in difference between involved and uninvolved FLC levels. If serum free light assay also unmeasurable, require at least 50% reduction in plasma cells, provided baseline was at least 30%
  * Very Good PR (VGPR) = Serum and urine M-protein detectable by immunofixation but not on electrophoresis, or >90% reduction in serum M-protein plus urine M-protein level <100 mg/24 h
Time Frame: up to 8 months
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab and Ixazomib
Number analyzed (Participants) | 2
percentage of participants | 0

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the time from starting study treatment to disease progression or death from any cause. The International Myeloma Working Group (IMWG) criteria defines progressive disease (PD) as at least 25% increase from lowest response value of any of the following:
  * Serum M-component (absolute increase must be at least 0.5 g/dL)
  * Urine M-component (absolute increase must be at least 200 mg/24 h)
  * If serum and urine M-protein unmeasurable, absolute increase in free light chain (FLC) must be >10 mg/dL. If FLC levels also unmeasurable, absolute increase in bone marrow plasma cell percentage must be at least 10%.
  * Definite development of new bone lesions or soft tissue plasmacytomas, or definite increase in size of existing bone lesions or soft tissue plasmacytomas
  * Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the plasma cell proliferative disorder
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab and Ixazomib
Number analyzed (Participants) | 2
months | 3.96 [1.15 to NA] — Upper limit was not reached due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Nivolumab and Ixazomib
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab and Ixazomib (N=2)
Constipation (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Personality change (mood changes) (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT04119336/Prot_SAP_000.pdf